CLINICAL TRIAL: NCT00813748
Title: Pharmacosurveillance Data Repository of Patients With and Without History of Anaphylactic Reactions Subsequent to Xolair(R) Dosing
Brief Title: Pharmacosurveillance Data Repository of Patients With and Without History of Anaphylactic Reactions Subsequent to Xolair Dosing
Acronym: X-PAND
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Q4458g
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Allergic Asthma
Keywords: Asthma; Anaphylaxis
MeSH Terms: conditions — Asthma; Anaphylaxis | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood

INTERVENTIONS:
Drug: Xolair

SUMMARY:
This study will establish a clinical data and serum repository of anaphylaxis cases associated with Xolair administration and control patients who have received Xolair without associated anaphylaxis. This is an observational repository and not an investigational clinical trial. Associated with the repository is an optional skin testing substudy.

ELIGIBILITY:
Inclusion Criteria for Cases:

* Confirmed anaphylaxis based on Sampson criteria subsequent to Xolair

Inclusion Criteria for Controls:

* At least 1 patient control among 4 controls who discontinued Xolair for at least 16 weeks but not more than 18 months at enrollment
* At least one dose of Xolair in the 18 months before the date of the case event (index date)
* No prior anaphylaxis or other hypersensitivity reaction subsequent to Xolair dosing, including any reactions to its components

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdelkader Rahmaoui, M.D., Study Director — Genentech, Inc.
Locations (7):
- United States (7):
  - Investigational Site, Los Angeles, California
  - Investigational Site, Valrico, Florida
  - Investigational Site, Hinsdale, Illinois
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, New York, New York
  - Investigational Site, Blue Bell, Pennsylvania
  - Investigational Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab Cases: Participants who received omalizumab (Xolair) and had anaphylaxis and/or severe hypersensitivity reactions which were adjudicated by an independent clinical expert to determine that they qualified as anaphylaxis or anaphylactoid reactions on the basis of the Sampson Criteria.
- Omalizumab Controls: Participants who received omalizumab within 18 months (either before or after) of the matched case participant's anaphylaxis occurrence (index date) and had not experienced anaphylaxis and/or severe hypersensitivity reactions subsequent to omalizumab dosing and were from the same site or region for their matched anaphylaxis case participant.
Period: Main Observational Study
Arm/Group | Omalizumab Cases | Omalizumab Controls
Started | 30 | 88
Completed | 30 | 88
Not Completed | 0 | 0
Period: Skin Test Substudy
Arm/Group | Omalizumab Cases | Omalizumab Controls
Started | 3 (Included participants who discontinued omalizumab for at least 16 weeks but not more than 18 months.) | 8 (Included participants who discontinued omalizumab for at least 16 weeks but not more than 18 months.)
Completed | 3 | 7
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Omalizumab Cases: Participants who received omalizumab and had anaphylaxis and/or severe hypersensitivity reactions which were adjudicated by an independent clinical expert to determine that they qualified as anaphylaxis or anaphylactoid reactions on the basis of the Sampson Criteria.
- Total: Total of all reporting groups
Arm/Group | Omalizumab Cases | Omalizumab Controls | Total
Number analyzed (Participants) | 30 | 88 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] — For Cases, age reported is the age at the time of the adjudicated event. For Controls, age reported is the age at the time of the adjudicated event experienced by the matched Case participant.
  years | 42.7 (16.41) | 45.4 (15.40) | 44.7 (15.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 60 | 87
  Male | 3 | 28 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Signs and Symptoms of Adjudicated Anaphylaxis Events - Case Participants
Description: Clinical signs and symptoms of adjudicated anaphylaxis events included: Cutaneous/Subcutaneous/Mucosal, Respiratory (R), Cardiovascular (CV), and Gastrointestinal (GIT) signs and symptoms.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants
  Cutaneous/Subcutaneous/Mucosal + R | 24
  Cutaneous/Subcutaneous/Mucosal + R + CV | 2
  Cutaneous/Subcutaneous/Mucosal + R + GIT | 1
  Cutaneous/Subcutaneous/Mucosal + CV | 1
  R + CV + GIT | 1
  CV | 1

2. Primary Outcome: Time From Last Omalizumab Dose to Adjudicated Anaphylactic Symptoms - Case Participants
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants. Here, number of participants analyzed signifies participants with available data for this outcome.
Measure: Median (Full Range); unit: minutes
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 27
minutes | 30 [0 to 210]

3. Primary Outcome: Categorical Time From Last Omalizumab Dose to Adjudicated Anaphylactic Symptoms - Case Participants
Description: Time from last omalizumab dose to adjudicated anaphylactic symptoms was classified as: less than (<) 30 minutes, 30-60 minutes, greater than (>) 60-90 minutes, >90-120 minutes, >120 minutes to 360 minutes, and missing. Number of participants in each time category is reported.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants
  <30 minutes | 13
  30-60 minutes | 8
  >60-90 minutes | 3
  >90-120 minutes | 2
  >120-360 minutes | 1
  Missing | 3

4. Primary Outcome: Total Omalizumab Doses Received When Adjudicated Anaphylactic Event Occurred - Case Participants
Description: Omalizumab doses were classified as: 1 dose, 2 doses, 3 doses, 4-20 doses, 21-40 doses, 41-60 doses, >60 doses, and missing. Number of participants in each dose category is reported.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants
  1 Dose | 6
  2 Doses | 3
  3 Doses | 2
  4-20 Doses | 8
  21-40 Doses | 4
  41-60 Doses | 4
  >60 Doses | 1
  Missing | 2

5. Primary Outcome: Treatment Received Following Adjudicated Anaphylactic Event - Case Participants
Description: Treatment received following adjudicated anaphylactic event was classified as: antihistamine, epinephrine, inhaled beta agonists, systemic corticosteroids, and other. Number of participants in each treatment category is reported. Participants could have received more than 1 treatment.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants
  Antihistamine | 23
  Epinephrine | 21
  Inhaled Beta Agonists | 13
  Systemic Corticosteroids | 19
  Other | 6

6. Primary Outcome: Outcome Attributed to Adjudicated Anaphylactic Event - Case Participants
Description: Outcomes of adjudicated anaphylactic event were classified as: death, life-threatening, required in-patient hospitalization or its prolongation, disabling, congenital anomaly/birth defect in offspring of participant, and other (outcome did not meet any of the above criteria, but may jeopardize the participant, and may require medical or surgical intervention to prevent one of the outcomes listed above). Number of participants in each outcome category is reported. Only outcomes with results are reported.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants
  Life-Threatening | 12
  In-Patient Hospitalization or its Prolongation | 6
  Other | 12

7. Primary Outcome: Number of Participants Reinitiating Omalizumab After Adjudicated Anaphylactic Event - Case Participants
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants | 4

8. Primary Outcome: Number of Participants With Prior Unadjudicated Anaphylactic Events - Case Participants
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants | 7

9. Primary Outcome: Treatment Following Prior Unadjudicated Anaphylactic Events - Case Participants
Description: Treatment received following prior unadjudicated anaphylactic events was classified as: antihistamine, epinephrine, inhaled beta agonists, systemic corticosteroids, and other. Number of participants in each treatment category is reported. Participants could have received more than 1 treatment.
Time Frame: Baseline (Enrollment Visit)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 5
participants
  Antihistamine | 4
  Epinephrine | 2
  Inhaled Beta Agonists | 3
  Systemic Corticosteroids | 1
  Other | 1

10. Primary Outcome: Number of Participants With Subsequent Unadjudicated Anaphylactic Events - Case Participants
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants | 3

11. Primary Outcome: Treatment Following Subsequent Unadjudicated Anaphylactic Events - Case Participants
Description: Treatment received following subsequent unadjudicated anaphylactic event was classified as: antihistamine, epinephrine, inhaled beta agonists, systemic corticosteroids, and other. Number of participants in each treatment category is reported. Participants could have received more than 1 treatment.
Time Frame: Baseline (Enrollment Visit)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 3
participants
  Antihistamine | 1
  Epinephrine | 1
  Inhaled Beta Agonists | 1
  Systemic Corticosteroids | 1
  Other | 1

12. Primary Outcome: Medications Received Within Two Weeks Prior to the Adjudicated Anaphylactic Event - Case Participants
Description: Number of participants in each medication class is reported. Participants could have received more than 1 medication class. NEC: Not Elsewhere Classified.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases
Number analyzed (Participants) | 30
participants
  5-Hydroxytryptamine Receptor 1 (5-HT1) Agonists | 1
  Adrenergics/Sympathomimetics | 3
  Aminoglycoside Antimicrobials | 1
  Analgesic/Other Drug Combinations | 2
  Analgesics | 4
  Angiotensin II Receptor Antagonists | 2
  Antacids NEC | 1
  Antianxiety Agents | 1
  Antidepressants NEC | 1
  Antidiuretics | 1
  Antiemetics NEC | 2
  Antihistamines | 16
  Antipsychotic and Antimanic Agents | 2
  Benzodiazepines | 6
  Biguanides | 1
  Bisphosphonates | 1
  Bronchodilators and Antiasthmatics | 29
  Calcium Channel Blocking Agents | 3
  Cephalosporin Antibiotics | 1
  Cough Preparations | 2
  Diuretics NEC | 1
  Glycopeptide Antibiotics | 1
  Herbal,Homeopathic,& Dietary Supplements | 1
  Histamine H2-receptor Antagonists | 3
  Laxatives and Stool Softeners | 1
  Leukotriene Receptor Antagonists | 21
  Macrolide Antibiotics | 2
  Miscellaneous Gastrointestinal Agents | 1
  Muscle Relaxants | 1
  Non-steroidal Anti-inflammatories | 2
  Opioid Analgesics | 1
  Penicillins | 1
  Peripheral and Cerebral Vascular Agents | 1
  Proton Pump Inhibitors | 10
  Salicylates | 1
  Sedatives and Hypnotics | 1
  Selective Serotonin Re-uptake Inhibitors | 4
  Sex Hormones | 3
  Statins | 2
  Steroid/Other Drug Combinations | 1
  Steroids | 22
  Supplements | 2
  Thiazide Diuretics | 1
  Thyroid Hormones | 4
  Tricyclic Antidepressants | 4
  Vitamins and Minerals | 2

13. Primary Outcome: Medications Within Two Weeks Prior to Blood Draw
Description: Number of participants in each medication class is reported. Participants could have received more than 1 medication class.
Time Frame: Baseline (Enrollment Visit)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases | Omalizumab Controls
Number analyzed (Participants) | 30 | 88
participants
  5-HT1 Agonists | 0 | 2
  5-Hydroxytryptamine Receptor 3 (5-HT3) Antagonists | 1 | 0
  Adrenergics/Sympathomimetics | 2 | 0
  Alpha-adrenoreceptor Antagonists | 2 | 4
  Aminoglycoside Antimicrobials | 0 | 1
  Aminosalicylates | 0 | 1
  Analgesic/Other Drug Combinations | 3 | 5
  Analgesics | 5 | 11
  Androgens and Anabolic Steroids | 0 | 3
  Angiotensin II Receptor Antagonists | 5 | 6
  Angiotensin-converting Enzyme Inhibitors | 1 | 6
  Anorexiants and CNS Stimulants | 2 | 6
  Antacids NEC | 0 | 1
  Antiallergic Agents NEC | 0 | 1
  Antiandrogens | 0 | 2
  Antianemic Agents | 0 | 2
  Antianginal Agents NEC | 0 | 1
  Antianxiety Agents | 1 | 2
  Anticoagulants | 0 | 4
  Anticonvulsants NEC | 3 | 12
  Antidepressants NEC | 1 | 10
  Antidiuretics | 1 | 0
  Antiemetics NEC | 2 | 4
  Antifungal Agents | 0 | 1
  Antiglaucoma Agents | 0 | 1
  Antigout Agents | 0 | 5
  Antihistamines | 19 | 57
  Antihypertensive Agents NEC | 2 | 9
  Antimalarial Agents | 0 | 1
  Antimetabolites | 0 | 2
  Antimicrobial/Other Drug Combinations | 0 | 1
  Antiparkinsonism Agents NEC | 0 | 1
  Antipsychotic and Antimanic Agents | 3 | 3
  Antispasmodics and Anticholinergics | 5 | 1
  Antitrichomonal Agents | 1 | 1
  Antiviral Agents NEC | 0 | 1
  Benzodiazepines | 9 | 10
  Beta-adrenoceptor Blocking Agents | 2 | 4
  Biguanides | 1 | 5
  Bisphosphonates | 1 | 3
  Bronchodilators and Antiasthmatics | 27 | 70
  Calcium Channel Blocking Agents | 6 | 12
  Calcium Compounds and Regulators | 4 | 7
  Cephalosporin Antibiotics | 0 | 1
  Cold and Sinus Remedies | 1 | 3
  Cough Preparations | 0 | 5
  Cox-2 Inhibitors | 1 | 2
  Dermatologic Agents | 1 | 2
  Diuretics NEC | 0 | 6
  Dopaminergic Agents | 2 | 0
  Enzymes | 0 | 1
  Fibrates | 0 | 2
  Folic Acid and Derivatives | 1 | 2
  Herbal,Homeopathic,& Dietary Supplements | 4 | 16
  Histamine H2-receptor Antagonists | 5 | 6
  Hypertensives | 1 | 0
  Hypoglycemics NEC | 1 | 3
  Immunosuppressants | 1 | 2
  Insulins | 0 | 2
  Laxatives and Stool Softeners | 1 | 3
  Leukotriene Receptor Antagonists | 19 | 49
  Lipid Regulating Agents NEC | 0 | 2
  Local Anesthetics | 1 | 0
  Loop Diuretics | 2 | 9
  Macrolide Antibiotics | 3 | 2
  Miscellaneous Cardiovascular Agents | 0 | 1
  Miscellaneous Drugs | 0 | 1
  Mucosal Protectants | 1 | 0
  Muscle Relaxants | 2 | 6
  Nitrofurans | 0 | 1
  Non Drug Therapies | 1 | 1
  Non-steroidal Anti-inflammatories | 6 | 9
  Opioid Analgesics | 2 | 6
  Parasympathomimetics and Antimyasthenics | 1 | 0
  Penicillins | 1 | 2
  Peripheral and Cerebral Vascular Agents | 1 | 0
  Pharmaceutic Aids | 1 | 2
  Pharmacotherapeutic Class (ES) Not Known | 0 | 3
  Phenothiazines | 1 | 0
  Platelet Aggregation Inhibitors | 0 | 3
  Proton Pump Inhibitors | 13 | 36
  Quinolone Antibiotics | 0 | 3
  Salicylates | 4 | 12
  Sedatives and Hypnotics | 2 | 5
  Selective Serotonin Re-uptake Inhibitors | 8 | 15
  Sex Hormones | 8 | 14
  Statins | 3 | 20
  Steroid/Other Drug Combinations | 0 | 3
  Steroids | 24 | 53
  Sulfonylureas | 2 | 1
  Supplements | 1 | 12
  Tetracyclines | 1 | 0
  Therapeutic Gases | 2 | 2
  Thiazide Diuretics | 3 | 3
  Thiazolidinediones | 0 | 2
  Thyroid Hormones | 5 | 12
  Tricyclic Antidepressants | 3 | 4
  Vaccines, Toxoids and Serologic Agents | 1 | 1
  Vitamins and Minerals | 9 | 24

14. Primary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATA) - Main Study
Description: Participants with positive immunoglobulin G (IgG) ATA, negative IgG ATA, positive immunoglobulin E (IgE) ATA, and negative IgE ATA are reported.
Time Frame: Baseline (Enrollment Visit)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases | Omalizumab Controls
Number analyzed (Participants) | 21 | 10
participants
  Participants with Positive IgG ATA | 0 | 0
  Participants with Negative IgG ATA | 21 | 10
  Participants with Positive IgE ATA | 0 | 0
  Participants with Negative IgE ATA | 21 | 10

15. Primary Outcome: Number of Participants With Positive Skin Reaction After Skin Prick Test - Skin Testing Substudy
Time Frame: Substudy Day 1
Population: Skin test substudy: all enrolled participants. One participant discontinued prematurely from the skin test substudy before providing data and was excluded.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases | Omalizumab Controls
Number analyzed (Participants) | 3 | 7
participants | 0 | 2

16. Primary Outcome: Number of Participants With ATA - Skin Testing Substudy
Description: Participants with positive IgG ATA, negative IgG ATA, positive IgE ATA, and negative IgE ATA are reported.
Time Frame: Substudy Week 10
Population: Skin test substudy: all enrolled participants. Here, number of participants analyzed signifies participants with available data for this outcome.
Measure: Number; unit: participants
Arm/Group | Omalizumab Cases | Omalizumab Controls
Number analyzed (Participants) | 3 | 6
participants
  Participants with Positive IgG ATA | 0 | 0
  Participants with Negative IgG ATA | 3 | 6
  Participants with Positive IgE ATA | 0 | 0
  Participants with Negative IgE ATA | 3 | 6

ADVERSE EVENTS:
Time Frame: Main observational study: Baseline (enrollment visit); Skin test substudy: 10 weeks
Description: One participant discontinued prematurely from the skin test substudy before providing data and was excluded. The term non-systematic signifies that the adverse events (AEs) were collected in a non-systematic manner where in addition to scheduled assessments, voluntary AE reporting was also allowed.
Groups:
- Observational Study: Omalizumab Cases - With Anaphylaxis; Skin Test Substudy: Omalizumab Cases - With Anaphylaxis: Participants who received omalizumab and had anaphylaxis and/or severe hypersensitivity reactions which were adjudicated by an independent clinical expert to determine that they qualified as anaphylaxis or anaphylactoid reactions on the basis of the Sampson Criteria.
- Observational Study: Omalizumab Controls - Without Anaphylaxis; Skin Test Substudy: Omalizumab Controls - Without Anaphylaxis: Participants who received omalizumab within 18 months (either before or after) of the matched case participant's anaphylaxis occurrence (index date) and had not experienced anaphylaxis and/or severe hypersensitivity reactions and were from the same site or region for their matched anaphylaxis case participant.
Arm/Group | Observational Study: Omalizumab Cases - With Anaphylaxis | Observational Study: Omalizumab Controls - Without Anaphylaxis | Skin Test Substudy: Omalizumab Cases - With Anaphylaxis | Skin Test Substudy: Omalizumab Controls - Without Anaphylaxis
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/88 | 1/3 | 0/7
Other Adverse Events (participants affected / at risk) | 0/30 | 0/88 | 1/3 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observational Study: Omalizumab Cases - With Anaphylaxis (N=30) | Observational Study: Omalizumab Controls - Without Anaphylaxis (N=88) | Skin Test Substudy: Omalizumab Cases - With Anaphylaxis (N=3) | Skin Test Substudy: Omalizumab Controls - Without Anaphylaxis (N=7)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — As per sponsor assessment this was a potential anaphylaxis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observational Study: Omalizumab Cases - With Anaphylaxis (N=30) | Observational Study: Omalizumab Controls - Without Anaphylaxis (N=88) | Skin Test Substudy: Omalizumab Cases - With Anaphylaxis (N=3) | Skin Test Substudy: Omalizumab Controls - Without Anaphylaxis (N=7)
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Endpoint prioritization was not specified in study protocol; hence, all endpoints are reported as primary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.